CLINICAL TRIAL: NCT01764230
Title: Prevention of Ovarian Function Damage by a GnRH Analogue During Chemotherapy in Hodgkin Lymphoma Patients
Acronym: OVARONKO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masaryk University (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: Principal Investigator, Martin Huser, MD, PhD., Masaryk University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Masaryk University
Record Dates: First submitted 2012-12-30; First posted 2013-01-09 (Estimated); Last update posted 2013-01-09 (Estimated); Status verified 2013-01

CONDITIONS: Hodgkin Lymphoma; Hodgkin Disease
Keywords: Hodgkin lymphoma; Hodgkin disease
MeSH Terms: conditions — Hodgkin Disease | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- case group (Experimental): Throughout the course of chemotherapy, patients were administered triptorelin (Diphereline SR 3 mg, Ibsen) in the form of i.m. injections, always once a month and simultaneously with the chemotherapy.
  Interventions: Drug: triptorelin
- control group (No Intervention): no intervention

INTERVENTIONS:
Drug: triptorelin — Throughout the course of chemotherapy, patients were administered triptorelin (Diphereline SR 3 mg, Ibsen) in the form of i.m. injections, always once a month and simultaneously with the chemotherapy.
  Other Names: triptorelin (Diphereline SR 3 mg, Ibsen)
  Arms: case group

SUMMARY:
Chemotherapy as one of the basic modalities of oncology treatment often leaves permanent implications and among the most common is infertility as a result of irreversible gonadal damage. This project sets the primary target to verify the protective effect GnRH analogues administration to protect ovarian tissue during three different regimens of chemotherapy in patients with Hodgkin disease (HD) in reproductive age.

DETAILED DESCRIPTION:
During the first two years of the project duration the curative anti-tumorous combined treatment in fertile patients with Hodgkin disease diagnosis will be carried out. Patients are to be divided into three groups according to the clinical stage of the disease and treated with the three types of the chemotherapeutic regimens comparable with toxicity. Patients will receive GnRH analogues during the chemotherapy for the gonadal protection by the mechanism of foliculogenesis inhibition in pre-pubertal stage. At the end of successful treatment according to stated criteria the ovarian function of every patient will be repeatedly evaluated in relation with toxicity of chemotherapy used. These ovarian function results will be compared with control group of patients without gonadal protection, which reproductive functions will be evaluated according the same method.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Hodgkin lymphoma
* FSH and LH levels in peripheral blood below 15 IU/l
* fertile age from 18 to 35 years
* female
* presence of both ovaries

Exclusion Criteria:

* ovarian tumours or cysts over 40 mm in diameter

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2004-01; Primary Completion 2007-07 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Premature ovarian failure after chemotherapy | 6 months after the end of chemotherapy
  Premature ovarian failure defined as levels of FSH over 15 IU/l in peripheral blood.
Premature ovarian failure after chemotherapy | 12 months after the end of chemotherapy
  Premature ovarian failure defined as levels of FSH over 15 IU/l in peripheral blood.

SECONDARY OUTCOMES:
Rate of premature ovarian failure according to the degree of toxicity of the chemotherapeutic regimen | 6 months after the end of chemotherapy
  A - ABVD 4x Adriamycin, bleomycin, vinblastin and dacarbazin
  B Combination of ABVD and BEACOPP regimens 4x Adriamycin, bleomycin, vinblastin and dacarbazinþbleomycin, etoposide, adriamycin, cyclophosphamide, vincristine, procarbazine and prednisone
  C BEACOPP regimen 8x - Bleomycin, etoposide, adriamycin, cyclophosphamide, vincristine, procarbazine and prednisone
Rate of premature ovarian failure according to the degree of toxicity of the chemotherapeutic regimen | 12 month after chemotherapy
  A - ABVD 4x Adriamycin, bleomycin, vinblastin and dacarbazin
  B Combination of ABVD and BEACOPP regimens 4x Adriamycin, bleomycin, vinblastin and dacarbazinþbleomycin, etoposide, adriamycin, cyclophosphamide, vincristine, procarbazine and prednisone
  C BEACOPP regimen 8x - Bleomycin, etoposide, adriamycin, cyclophosphamide, vincristine, procarbazine and prednisone

CONTACTS AND LOCATIONS:
Overall Officials: Martin Huser, MD, PhD, Principal Investigator — Masaryk University
Locations (1):
- Brno University Hospital and Masaryk University School of Medicine, Brno, Czechia

REFERENCES:
- [Result] Huser M, Crha I, Ventruba P, Hudecek R, Zakova J, Smardova L, Kral Z, Jarkovsky J. Prevention of ovarian function damage by a GnRH analogue during chemotherapy in Hodgkin lymphoma patients. Hum Reprod. 2008 Apr;23(4):863-8. doi: 10.1093/humrep/den005. Epub 2008 Feb 7. PMID 18258763